CLINICAL TRIAL: NCT06543823
Title: The Use of Suprathel®250 as a Novel Therapeutical Option for Mucosal Healing in Head and Neck Surgery
Brief Title: ST250 as a Therapeutic Option for Head & Neck Reconstruction
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alaa Emara (Other)
Responsible Party: Sponsor-Investigator, Alaa Emara, Associate Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ST250 mucosal application
Record Dates: First submitted 2024-07-31; First posted 2024-08-09 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-01

CONDITIONS: Tonsillitis
Keywords: PLA membrane; Biodegradable membrane; Synthetic; Tonsillectomy
MeSH Terms: conditions — Tonsillitis

STUDY DESIGN:
Intervention Model Description: An interventional group with the application of the SupraTHEL 250 membrane and the control group with no membrane applied on the wound bed
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Sham Comparator): The wound bed is left bare after the tonsillectomy procedure
  Interventions: Other: Comparator
- SupraTHEL 250 group (Experimental): The SupraTHEL 250 membrane is suture ionto the wound bed after the tonsillectomy procedure
  Interventions: Device: SupraTHEL 250

INTERVENTIONS:
Device: SupraTHEL 250 — the membrane is placed onto the wound bed and fixed in place by resorbable interrupted sutures
  Arms: SupraTHEL 250 group
Other: Comparator — no membrane is placed onto the wound bed , left bare to heal
  Arms: Study group

SUMMARY:
To assess the use of SupraThel 250 for mucosal reconstruction in the Head & Neck region. The membrane will be applied after tonsillectomy procedures and compared to bare wounds' healing

DETAILED DESCRIPTION:
After tonsillectomy procedures, the wound is usually left bare to heal. This causes severe pain postoperatively and postoperative hemorrhage. SupraTHEL 250 is a synthetic biodegradable PLA membrane which is proven as a skin membrane in burn wounds with excellent result. We therefore hypothesize that the use opf SupraTHEL 250 after tonsillectomy procedures will allow for faster , less painful healing of the wound bed which allows for a better quality of life for the patients.

ELIGIBILITY:
Inclusion Criteria:

* recurrent episodes of tonsillar infection

Exclusion Criteria:

* children
* pregnant/ breastfeeding women
* patients undergoing chemo / radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pain scores | upto 5 days postoperatively
  Visual Analogue Scores (0-10; 0 lowest , 10 highest)

SECONDARY OUTCOMES:
Quality of Life , Tonsillectomy Outcome Inventory - 14 | 5 days Postoperative
  assessment of patients quality of life according to a set of questions

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Emara, Principal Investigator — Cairo University
Locations (1):
- MarienHospital, Stuttgart, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No